CLINICAL TRIAL: NCT05271578
Title: MRI and Biological Markers of Acute E-Cigarette Exposure in Smokers and Vapers
Acronym: AeCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 850432; R01HL155243 (NIH)
Record Dates: First submitted 2022-01-20; First posted 2022-03-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Vascular Reactivity; Serum Biomarkers
Keywords: Magnetic Resonance Imaging; Electronic Cigarettes; Endothelial Dysfunction; Nicotine; Inflammation
MeSH Terms: conditions — Vaping; Inflammation

STUDY DESIGN:
Intervention Model Description: The study will be conducted in a three-period crossover design and will involve active e-cig (electronic cigarette) and tobacco cigarette users undergoing three different interventions (blinded to the investigators).
  The three periods will consist of (1) electronic cigarette vaping without nicotine, (2) electronic cigarette vaping with nicotine, (3) tobacco cigarette smoking. Sequence order will be established by means of a computer-generated randomization scheme.
Who Masked: Participant, Investigator
Masking Description: Blinding to nicotine and placebo containing standardized electronic research cigarettes and standardized tobacco research cigarettes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers (Experimental): Conventional tobacco cigarette smokers
  Interventions: Device: Standardized Electronic Research Cigarette; Device: Nicotine Research Cigarette
- Vapers (Experimental): Electronic cigarette vapers
  Interventions: Device: Standardized Electronic Research Cigarette; Device: Nicotine Research Cigarette

INTERVENTIONS:
Device: Standardized Electronic Research Cigarette — Standardized Research Electronic Cigarette Device, Standardized Research Electronic Cigarette Tobacco 5%, Standardized Research Electronic Cigarette Tobacco (placebo) 0% (NJOY, LLC, Tobacco Product Master File #STN MF0000274)
  Other Names: SREC
Device: Nicotine Research Cigarette — Conventional Nicotine Tobacco Cigarette (National Institute of Drug Abuse, Drug Supply Program, Tobacco Product Master File #NRC600)
  Other Names: NRC

SUMMARY:
To examine vascular reactivity and inflammatory biomarkers via quantitative magnetic resonance imaging (MRI) and blood serum, respectively, in a crossover study where active vapers (electronic cigarette users) and smokers will undergo three separate acute exposure-episodes of electronic cigarette +/- nicotine and tobacco-cig. The MRI exams and blood draws will be performed pre- and post-exposure. The results will be compared against baseline values derived from a group of non-smokers/non-vapers, who will also undergo a blood draw and MRI.

DETAILED DESCRIPTION:
This work is an extension of prior funded work on the acute effects of nicotine free electronic cigarette aerosol on vascular function and inflammatory biomarkers in healthy non-smokers. Here, the investigators will examine vascular reactivity and inflammatory biomarkers using quantitative magnetic resonance imagine (MRI) and blood serum in a crossover study, with active vapers (electronic cigarette users) and smokers undergoing three, separate-day, acute exposure-episodes of smoking a tobacco cigarette, an electronic cigarette without nicotine, and an electronic cigarette with nicotine. Participants will undergo an MRI exam and a blood draw pre- and post-exposure-episode.

The investigators hypothesize that all three paradigms will cause a transient response but greatest for tobacco and nicotinized electronic cigarettes. The results will be compared against baseline values derived from a group of non-smokers/non-vapers, who will undergo a blood draw and MRI only. Eligible participants will be healthy, males and females, current, habitual users of electronic or tobacco cigarettes (except for the non-smoking/non-vaping comparison group), 21 to 45 years of age, and without co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5 to 30
* Current users of electronic cigarettes or tobacco cigarettes with a use history of six months or greater.

Exclusion Criteria:

* Cancer
* HIV
* Mental illness in which the participant is not of proper cognizance
* Overt cardio- or neurovascular disease (prior heart attack, stroke, transient ischemic attacks)
* Serious arrhythmias
* Bronchospastic disease
* Upper respiratory tract infection within the past six weeks
* Medication affecting vascular function
* Antibiotics
* Magnetic resonance imaging contraindications (metallic implants/intraocular foreign bodies, claustrophobia, cardiac/cochlear implantable electronic devices, etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Changes in magnetic resonance imaging (MRI) biomarkers of endothelial dysfunction: aortic arch | Pre-Inhalation (baseline) to post-inhalation (60 minutes)
  Changes in stiffness of aortic arch in terms of pulse-wave velocity measured in meters per second.
Changes in magnetic resonance imaging (MRI) biomarkers of endothelial dysfunction: cerebral vascular reactivity | Pre-Inhalation (baseline) to post-inhalation (60 minutes)
  Rate of change in the blood flow velocity [centimeters per second (squared)] in a major draining vein in response to volitional apnea.
Changes in magnetic resonance imaging (MRI) biomarkers of endothelial dysfunction: femoral artery flow-mediated dilation | Pre-Inhalation (baseline) to post-inhalation (60 minutes)
  Percentage measure of the change of a cross-sectional area of the superficial femoral artery.
Changes in magnetic resonance imaging (MRI) biomarkers of endothelial dysfunction: venous oxygen saturation | Pre-Inhalation (baseline) to post-inhalation (60 minutes)
  Assessment of microvascular function by monitoring the changes in tissue blood oxygenation measured in percentage in response to a cuff-induced ischemia.
Changes in magnetic resonance imaging (MRI) biomarkers of endothelial dysfunction: blood flow velocity | Pre-Inhalation (baseline) to post-inhalation (60 minutes)
  Macrovascular function is evaluated by monitoring hyperemia in response to a cuff-induced ischemia by measuring femoral artery blood flow velocity in centimeters per second.
Changes in blood inflammatory biomarkers | Pre-Inhalation (baseline) to post-inhalation (60 minutes)
  Measured in nanograms/milliliter of plasma, the following biomarkers are collectively associated with damage to blood vessels and recruitment of immune cells into the vascular tissue leading to severe oxidative stress and tissue damage in the vasculature: biomarker of oxidative stress (c-reactive protein) and biomarkers of inflammation (NLR family pyrin domain containing 3, damage-associated molecular pattern protein HMGB1, tumor necrosis factor alpha, interleukin 1β, interleukin 18, interferon gamma, monocyte chemoattractant protein, and macrophage inflammatory protein).

CONTACTS AND LOCATIONS:
Overall Officials: Felix W Wehrli, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No